CLINICAL TRIAL: NCT00200317
Title: Interactive Technologies to Increase Exercise Behavior
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: University of Pittsburgh (Other); Brown University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01HL069866 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2005-09

CONDITIONS: Cardiovascular Disease
Keywords: Exercise; Internet; Print; Randomized Controlled Trial; Exercise Intervention
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

INTERVENTIONS:
Behavioral: Internet and print-based interventions

SUMMARY:
The purpose of this study is to examine if an individually tailored Internet intervention is more efficacious than an individually tailored print-based intervention and standard Internet intervention for physical activity adoption and maintenance among sedentary adults.

DETAILED DESCRIPTION:
As many as 75% of Americans do not engage in regular physical activity and 25% are completely inactive. The risk of cardiovascular disease is almost doubled among people who are physically inactive, comparable to the risk associated with increased systolic blood pressure, cigarette smoking, and elevated serum cholesterol. To make an impact on physical activity prevalence at the population level, research must focus at the interface between clinical efficacy trials and large-scale dissemination studies. Studies at this interface must compare proven interventions with new innovations that have the potential to reach large numbers of sedentary Americans.

The objective of this study is to determine the differential effect of intervention delivery channel (Tailored Internet versus Tailored Print) on physical activity adoption and maintenance in previously sedentary adults. To our knowledge, no studies have examined the efficacy of a Tailored Internet-based physical activity intervention. Thus, we will conduct a randomized controlled clinical trial comparing three groups, 1) Internet-based motivationally-tailored individualized feedback (Tailored Internet); 2) print-based motivationally-tailored individualized feedback which has previously shown to be efficacious (Tailored Print); and 3) websites currently available to the public (Standard Internet comparison group). Two hundred and forty healthy, sedentary women and men ages 18-65 will be randomly assigned to one of the three groups. The Tailored Internet and Tailored Print arms will be matched on frequency and content of contact. Data will be collected at baseline, 6, and 12 months using well-established physical activity and physical performance measures, as well as a comprehensive set of psychosocial questionnaires. Our primary hypothesis is that individuals randomized to the Tailored Internet arm will exhibit significantly higher levels of physical activity participation at 6 and 12 months than individuals in the Tailored Print arm due to the enhanced capabilities of the Internet (e.g., immediacy of feedback and enhanced graphics). And, in addition, subjects randomized to the Tailored Internet or Tailored Print conditions will exhibit significantly higher levels of physical activity participation at 6 and 12 months than those in the Standard Internet comparison condition. Other questions of interest will include an examination of potential moderators and mediators of the intervention-physical activity relationship. This study will contribute important information regarding the relative efficacy of Internet and print-based interventions, each of which can be utilized for widespread public health dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary, defined as exercising less than 90 minutes per week
* Lack of access to the Internet
* Lack of access to receiving mail

Exclusion Criteria:

* Coronary heart disease (history of myocardial infarction or symptoms of angina)
* Diabetes
* Stroke
* Osteoarthritis
* Osteoporosis
* Orthopedic problems which would limit treadmill testing
* Other medical or psychological problems that could make adherence with the study protocol difficult or dangerous
* Consumption of three or more alcoholics drinks per day
* Current or planned pregnancy
* Planning to move from the area within the next year
* Current suicidal ideation or psychosis
* Current clinical depression
* Recent hospitalization due to a psychiatric disorder
* Taking medication that may impair physical activity tolerance or performance (e.g., beta blockers).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2003-02; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Minutes of physical activity per week based on 7-Day Physical Activity Recall Interview.

SECONDARY OUTCOMES:
Minutes of physical activity per week based on objective physical activity monitor (ActiGraph);
Minutes of walking on a treadmill; and Estimated Vo2 on treadmill test.

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, Ph.D., Principal Investigator — Brown Medical School & The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Marcus BH, Lewis BA, Williams DM, Dunsiger S, Jakicic JM, Whiteley JA, Albrecht AE, Napolitano MA, Bock BC, Tate DF, Sciamanna CN, Parisi AF. A comparison of Internet and print-based physical activity interventions. Arch Intern Med. 2007 May 14;167(9):944-9. doi: 10.1001/archinte.167.9.944. PMID 17502536